CLINICAL TRIAL: NCT03804671
Title: Investigation of Pharmacokinetics and Absolute Oral Bioavailability of BI 730357 Administered as an Oral Dose With an Intravenous Microtracer Dose of BI 730357 BS (C-14) in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Measure the Amount of BI 730357 in the Blood When Taken as a Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1407-0033; 2018-003103-19 (EudraCT Number)
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): Test treatment T followed by Reference treatment R
  Interventions: Drug: BI 730357; Drug: BI 730357 mixed with [C-14] BI 730357 BS

INTERVENTIONS:
Drug: BI 730357 — Oral dose
Drug: BI 730357 mixed with [C-14] BI 730357 BS — Intravenous dose

SUMMARY:
To investigate the absolute oral bioavailability of BI 730357 administered as tablet compared with [C-14]BI 730357 BS administered as intravenous microtracer

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Further inclusion criteria apply

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 139 mmHg, diastolic blood pressure outside the range of 45 to 89 mmHg, or pulse rate outside the range of 40 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Clinically significant gastrointestinal (including known or suspected inflammatory bowel disease), hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Ooi QX, Kristoffersson A, Korell J, Flack M, L Plan E, Weber B. Bounded integer model-based analysis of psoriasis area and severity index in patients with moderate-to-severe plaque psoriasis receiving BI 730357. CPT Pharmacometrics Syst Pharmacol. 2023 Jun;12(6):758-769. doi: 10.1002/psp4.12948. Epub 2023 May 1. PMID 36919398
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed as a non-randomised, open-label, single arm, single period trial design in healthy male subjects in order to investigate the absolute oral bioavailability compared to the intravenous administered reference treatment of BI 730357.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- All Subjects: 1 tablet with 50 milligram (mg) BI 730357 was administered as a single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as test treatment (T) followed by 100 microgram (μg) of BI 730357 base (BS) (C-14) (2 μg radiolabelled [C-14]BI 730357 BS mixed with 98 μg unlabeled BI 730357) administered as 15 minutes (min) intravenous (i.v.) infusion as reference treatment (R) starting 1.25 hours (h) after oral administration.
Period: Overall Study
Arm/Group | All Subjects
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Treated set (TS) included all subjects who received at least 1 dose of trial medication. All 6 subjects were included in the TS. The safety analysis and the presentation of demographic and baseline characteristics were based on the TS.
Arm/Group | All Subjects
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 730357 Over the Time Interval From 0 to Infinity (Dose Normalized).
Description: Area under the concentration-time curve of the analyte over the time interval from 0 to infinity (AUC0-∞). For both arms results are presented in millimole (mmol) * hours (h) / Litre (L) / kilogram (kg). This was achieved by transforming the reference arm to the treatment arm and normalizing the results according to the respective dose.
Time Frame: Test treatment T: within 3h before and 1,1.5,2,2.5,3.5,5,7,12,24,72,120,168h after oral administration. Reference treatment R: within 3h before and 5,10,15,30,45 minutes and 1.25,2.25,3.75,5.75,10.75,22.75,70.75,118.75,166.75h after start of iv infusion.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least one pharmacokinetic (PK) endpoint that was defined as primary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: mmol*h/L/kg
Groups:
- BI 730357 50mg Tablet (T): 1 tablet with 50 milligram (mg) BI 730357 was administered as a single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as test treatment (T).
- BI 730357 BS (C-14) 100 µg Infusion (R): 100 microgram (μg) of BI 730357 BS (C-14) (2 μg radiolabelled [C-14]BI 730357 base (BS) mixed with 98 μg unlabelled BI 730357) administered as 15 minutes (min) intravenous (i.v.) infusion as reference treatment (R) starting 1.25 hours (h) after oral administration of test treatment (T).
Arm/Group | BI 730357 50mg Tablet (T) | BI 730357 BS (C-14) 100 µg Infusion (R)
Number analyzed (Participants) | 6 | 6
mmol*h/L/kg | NA (NA) — Geometric Mean is adjusted Geometric Mean = 160.38 Standard Error is Geometric standard error (gSE) = 1.16 | NA (NA) — Geometric Mean is adjusted Geometric Mean = 228.07 Standard Error is Geometric standard error (gSE) = 1.16
Statistical Analysis 1: Comparison: BI 730357 50mg Tablet (T) vs BI 730357 BS (C-14) 100 µg Infusion (R); Test type: Other — Absolute bioavailability. The statistical model was an ANOVA on the logarithmic scale including the fixed effect for 'formulation' and 'subject' as a random effect; Ratio of the geometric means (T/R) % = 70.32, 90% CI 2-sided [56.69 to 87.23] — The geometric coefficient of variation (gCV) = 18.7. Ratio was calculated as (AUC0-∞/dose) oral /(AUC0-∞/dose) intravenous multiplied by 100

ADVERSE EVENTS:
Time Frame: From the first administration of trial drug to the end of residual effect period up to 7 days.
Description: Adverse events are reported based on treated set (TS). This subject set included all subjects who were randomized and treated with at least 1 dose of trial drug. The TS was used for safety analyses.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=6)
Catheter site bruise (General disorders) | 1
Erection increased (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03804671/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT03804671/SAP_001.pdf